CLINICAL TRIAL: NCT05328141
Title: Measuring Dietary Iron Absorption From Edible Insects and Assessing the Effect of Chitin Content on Iron Bioavailability: Stable Iron Isotope Studies in Young Women (Study 2, Xylotrupes Gideon)
Brief Title: Measuring Dietary Iron Absorption From Edible Insects and Assessing the Effect of Chitin Content on Iron Bioavailability (Study 2)
Acronym: Sustironable2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Swiss Federal Institute of Technology (Other)
Collaborators: Zurich University of Applied Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: Sust-iron-able2
Record Dates: First submitted 2022-04-07; First posted 2022-04-14 (Actual); Last update posted 2022-06-10 (Actual); Status verified 2022-06

CONDITIONS: Iron-deficiency
Keywords: edible insects; iron bioavailability; ascorbic acid; Xylotrupes gideon
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — Bread; Butter; Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Bread and butter (Experimental): A toast bread with butter meal without insect biomass with FeSO4 (isotopic iron 54)
  Interventions: Other: Bread and butter
- X.gideon (Experimental): Intrinsically labelled (57Fe) or non labelled X.gideon flour mixed with butter and sugar meal with FeSO4 (extrinsic label, isotopic iron 58)
  Interventions: Other: X.gideon
- X.gideon with ascorbic acid (Experimental): Intrinsically labelled (57Fe) or non labelled X.gideon flour mixed with butter and sugar meal with FeSO4 (extrinsic label, isotopic iron 58) and ascorbic acid
  Interventions: Other: X.gideon with ascorbic acid

INTERVENTIONS:
Other: Bread and butter — A bread with butter meal without insect biomass with FeSO4 (isotopic iron 54)
  Arms: Bread and butter
Other: X.gideon — Intrinsically labelled (57Fe) or non labelled X.gideon flour mixed with butter and sugar meal with FeSO4 (extrinsic label, isotopic iron 58)
  Arms: X.gideon
Other: X.gideon with ascorbic acid — Intrinsically labelled (57Fe) or non labelled X.gideon flour mixed with butter and sugar meal with FeSO4 (extrinsic label, isotopic iron 58) and ascorbic acid
  Arms: X.gideon with ascorbic acid

SUMMARY:
Due to the growing world population, there is a need to develop viable ecological and nutritional alternatives to animal food products. However, animal products are a key dietary source of well-absorbed iron, and iron deficiency and iron deficiency anemia remain highly prevalent in high- and low-income countries. Meat and fish provide a substantial proportion of absorbed iron in the western diet by two distinct components: a) heme iron is well absorbed (20-45% fractional absorption) and is not affected by most dietary enhancers and inhibitors, which often affect non-heme iron absorption; b) peptides in muscle meat exert an enhancing effect the absorption of non-heme iron contained in other meal components. The potential of edible insects as a dietary source of well-absorbed iron has not been investigated in detail. In particular, it is unclear whether insects provide an iron moiety similar to hemoglobin which would be well absorbed and unaffected by other dietary components, and whether their presence in a test meal exerts an enhancing effect on iron bioavailability from the whole meal.

To differentiate iron absorption from insect biomass from other sources, insects will be intrinsically labelled with the stable iron isotope 57Fe, while other food iron components will be labelled with the iron isotope 58Fe.The present studiy will provide novel data to elucidate the nutritional value as sources of dietary iron of insect species Xylotrupes gideon. X. gideon is an insect species traditionally widely consumed in SubSaharan Africa and South East Asia and recognised by FAO as an edible insect species. X gideon is produced in ZHAW facilities in Linthal, Switzerland under controlled conditions aiming to a highly sustainable and high nutritional value food product. Furthermore the benefit of ascorbic acid addition to X.gideon biomass on iron absorption will be quantified.

ELIGIBILITY:
Inclusion Criteria:

* Female, 18 to 45 years old
* Normal Body Mass Index (18.5 - 25 kg/m2)
* Body weight ≤ 55 kg
* Non-anemic (hemoglobin (Hb) >12.0 g/dL)
* Serum Ferritin < 25 μg/L;
* Normal CRP (<5.0 mg/L), indicating no inflammation
* Knowledge of English at least at level B2 (assessed by self-declaration)
* Signed informed consent

Exclusion Criteria:

* Pregnancy (assessed by self-declaration)
* Lactating up to 6 weeks before study initiation
* Any metabolic, gastrointestinal kidney or chronic disease such as diabetes, hepatitis, hypertension, cancer or cardiovascular diseases (according to the participants own statement)
* Continuous/long-term use of medication (except for oral contraceptives and anti-acne medication)
* Consumption of mineral and vitamin supplements within 2 weeks prior to 1st meal administration
* Blood transfusion, blood donation or significant blood loss (accident, surgery) over the past 4 months
* Earlier participation in a study using iron stable isotopes or participation in any clinical study within the last 30 days
* Participant who cannot be expected to comply with study protocol (e.g. not available on certain study appointments
* Cigarette smoking ( > 1 cigarette per day)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Estimated)
Dates: Start 2022-05-20 (Actual); Primary Completion 2022-07-20 (Estimated); Study Completion 2022-07-30 (Estimated)

PRIMARY OUTCOMES:
Fractional Iron absorption | 30th day of the study
  Fractional iron absorption will be calculated based on the shift of the iron isotope ratios in the collected blood samples after the administration of the intervention products .Fractional iron absorption will be measured as erythrocyte incorporation of the naturally occurring iron forms with different masses used to label the iron supplements.

SECONDARY OUTCOMES:
Hemoglobin (Hb) | screening (-1), day 16th and day 30th of the study
  Iron status marker
Plasma ferritin (PF) | screening (-1), day 16th and day 30th of the study
  Iron status marker
C-Reactive Protein (CRP) | screening (-1), day 16th and day 30th of the study
  Inflammation status
Soluble transferring receptor (sTfR) | screening (-1), day 16th and day 30th of the study
  Iron status marker
Body iron stores (BIS) | screening (-1), day 16th and day 30th of the study
  Iron status marker
Alpha 1 acid glycoprotein (AGP) | screening (-1), day 16th and day 30th of the study
  Inflammation marker

CONTACTS AND LOCATIONS:
Overall Officials: Nikolin Hilaj, MSc, Principal Investigator — Laboratory of Human Nutrition ETH Zürich
Locations (1):
- ETH Zurich, Laboratory of Human Nutrition, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No